CLINICAL TRIAL: NCT05523596
Title: A Phase 1 Non-Randomized Open Label Study of ICM20
Brief Title: A Phase 1 Study of the Safety and Tolerability of ICM20 in Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IC-MedTech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ICM003
Record Dates: First submitted 2022-08-26; First posted 2022-08-31 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-07

CONDITIONS: Safety Issues
MeSH Terms: interventions — benzonidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 (Experimental): ICM20
  Interventions: Drug: ICM20
- Dose Level 2 (Experimental): ICM20 and benznidazole ascending dose 2
  Interventions: Drug: ICM20; Drug: Benznidazole
- Dose Level 3 (Experimental): ICM20 and benznidazole ascending dose 3
  Interventions: Drug: ICM20; Drug: Benznidazole
- Dose Level 4 (Experimental): ICM20 and benznidazole ascending dose 4
  Interventions: Drug: ICM20; Drug: Benznidazole

INTERVENTIONS:
Drug: ICM20 — small molecules
Drug: Benznidazole — small molecule
  Arms: Dose Level 2; Dose Level 3; Dose Level 4

SUMMARY:
A Phase 1 Non-Randomized Open Label Study of Oral ICM20

DETAILED DESCRIPTION:
This is a Phase 1 open label study to access the safety and tolerability of ICM20 alone and in combination with benznidazole

ELIGIBILITY:
Inclusion Criteria:

* ≥18 to 70 years of age
* ≥125 and ≤200 pounds
* Diagnosis of chagas documented by positive serology
* No prior chagas treatment
* Able to swallow capsules and tablets
* Laboratory values:

Blood: Hemoglobin ≥9; Polymorphonuclear white blood cells >1000; Platelets >50,000 Liver Function Tests ≤ 2 Times Upper Limit of Normal Serum Creatinine ≤2.0 Prothrombin time, partial thromboplastin time within normal limits HemoglobinA1C <7

* Human immunodeficiency virus negative
* Stable on current prescription medications
* Not pregnant, lactating, or planning to get pregnant
* Both men and women who are not surgically sterile, or post-menopausal, must agree to avoid pregnancy
* Willing to abstain from alcohol
* Able and willing to give informed consent

Exclusion Criteria:• Prior chagas treatment

* Known hypersensitivity to either study drug or its constituents
* Requires the continuing use of amiodarone, monoamine oxidase inhibitors, phenytoin, phenobarbital, disulfiram, anticoagulants or procoagulants, drugs or products containing alcohol or propylene glycol.
* Coagulopathy
* Glucose-6-phosphate dehydrogenase deficiency
* History, signs, or symptoms of heart failure
* History of heartburn, gastroesophageal reflux disease, or ulcers
* Unstable medical condition
* Immunodeficiency
* Requires surgery or surgical procedure within 90 days of Screening.
* Use of an investigational product within 56 days prior to baseline
* Unwilling to discontinue use of disallowed products
* Unable to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | through study completion, 90 days
  Number of participants with treatment related adverse events, based on a modified World Health Organization toxicity grading scale

SECONDARY OUTCOMES:
Percentage of participants on study drug at Day 28 and at Day 60 | 60 days
  Percentage of participants that are still taking the assigned study drug at Day 48 and at Day 60
Percentage of participants with a change from baseline in physical examination based on a review of systems | 90 days
  Percentage of participants that demonstrate a clinically relevant change from baseline on physical examination based on a review of systems
Percentage of participants with a change from baseline in vital signs (temperature in degrees Fahrenheit, respiratory rate in breaths per minute, heart rate in beats per minute, blood pressure in millimeters mercury) | 90 days
  Percentage of participants with a clinically relevant change from baseline in vital signs
Percentage of participants with a change from baseline in blood and urine tests | 90 days
  Percentage of participants that show a clinically relevant change from baseline
Percentage of participants with a change from baseline in the electrocardiogram | 90 days
  Percentage of participants that show a change in the twelve lead electrocardiogram

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Parkway Medical, Glen Burnie, Maryland
  - Baylor College of Medicine, Houston, Texas
  - Culmore Clinic, Falls Church, Virginia